CLINICAL TRIAL: NCT05309109
Title: Effect of Medium Cut-Off Hemodialysis on Protein Energy Wasting: The EMCOPEW Study. Medium Cut-Off Hemodialysis and Protein Energy Wasting
Brief Title: Effect of Medium Cut-Off Hemodialysis on Protein Energy Wasting: The EMCOPEW Study
Acronym: EMCOPEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EMCOPEW
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: hemodialysis; protein energy wasting; medium cut-off dialyzer; lean mass; bioimpedance
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MCO-HD group (Experimental): Hemodialysis sessions using the Theranova 500™ (Baxter healthcare Corporation Deerfield, USA; surface area 2 m², ultrafiltration coefficient: 59 ml/h/mmHg)
  Interventions: Other: Hemodialysis sessions
- HF-HD group (Experimental): Hemodialysis sessions using the Elisio 21H™ (Nipro Europe, Zaventen Belgium; surface area 2.1 m², ultrafiltration coefficient: 82 ml/h/mmHg)
  Interventions: Other: Hemodialysis sessions

INTERVENTIONS:
Other: Hemodialysis sessions — Patients will receive thrice weekly 4 hours hemodialysis sessions during 12 months.

SUMMARY:
In patients on maintenance hemodialysis (HD), protein energy wasting (PEW) defined as loss of muscle mass and fuel reserves of the body is frequent and associated with severe morbidity and mortality. Several factors, including inflammation, oxidative stress, metabolic disorders, loss of nutrients, diabetes, retention of middle molecule uremic toxins and dialysis procedure contribute to PEW. It has been previously reported that intensive HD treatments such as short daily and nocturnal HD may improve nutritional parameters. Moreover, post-dilution Online hemodiafiltration (OL-HDF) may also improve PEW by preserving lean body mass evaluated by bioimpedance analysis (BIA) probably through decreased inflammation, stimulation of appetite and better removal of uremic toxins. The recently developed medium cut-off dialyzer (MCO) in HD has demonstrated efficient depuration of middle uremic toxins as compared to high flux HD (HF-HD), similar to that of OL-HDF. Both MCO-HD and OL-HDF may exert beneficial effects on PEW, since they increase removal of higher weight middle molecules, which mostly encompass proteins related to inflammation and PEW in the uremic milieu

DETAILED DESCRIPTION:
In a previous randomized study, we found, that after 3 months, MCO-HD was associated with higher middle molecules removal and significant decrease in beta2-microglobulin, oxidized low-density lipoprotein, kappa and lambda free light chain pre-dialysis levels, without change in other inflammatory and oxidative stress biomarkers. In addition, compared to HF-HD, a modulation of inflammation has been demonstrated with MCO-HD in another randomized trial. After 3 months, MCO-HD was shown to downregulate the expression of the pro-inflammatory IL-6 and tumor necrosis factor (TNF) mRNA in peripheral leucocytes. Moreover, higher removal and decrease in TNF alpha level with concurrent reduced resistance to erythropoiesis stimulating agents (ESA) has been also reported with MCO-HD. However, the long-term effects of MCO-HD on inflammatory, uremic toxins and malnutrition biomarkers remain to be established.

To test the hypothesis that MCO-HD may positively affect body composition and nutritional status in HD patients we performed a 12-month single center retrospective pilot study. Compared to HF-HD, MCO-HD resulted in an improved variation rate of serum pre-dialysis creatinine level, lean tissue, skeletal muscle mass and index assessed by BIA, which are presumably good surrogate markers of PEW.

The aim of the present prospective, controlled randomized study is to evaluate the effect of MCO-HD on PEW, compared to standard HF-HD in chronic hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to give signed informed consent
* Age ≥ 18 years
* Patients established on HF-HD trice weekly four hour-sessions for at least 3 months.
* Patients able to walk
* Body mass index ≥ 20 and < 40 Kg/m2

Exclusion Criteria:

* Any uncontrolled medical condition, psychiatric disorder or biological abnormality that might interfere with subject's participation or ability to sign an informed consent.
* Implanted pace maker or cardioverter defibrillator
* Pregnant or breast-feeding women
* Active malignant disease, chronic inflammatory disease or other critical illnesses that may interfere with inflammatory parameters. Baseline C-reactive protein > 35 mg/l.
* Amputated limbs
* Prescription of oral or intra venous nutrition supplements
* Significant residual kidney function as defined by an urine output > 500 mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
The change from baseline to the end of the study in lean tissue mass measured using Bioimpedance analysis through the study. | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Poitiers, Poitiers
  - AURA Poitou-Charentes, Saint-Benoît

IPD SHARING:
Plan to Share IPD: No